CLINICAL TRIAL: NCT00464347
Title: Multi-Center, Randomized, Phase II Clinical Trial to Study the Effects of Preservative-Free Triamcinolone Acetonide and Avastin® in Combination With Photodynamic Therapy in Participants With Neovascular Age Related Macular Degeneration
Brief Title: TAC-PF, Avastin® in Combination With Photodynamic Therapy to Treat Age Related Macular Degeneration
Acronym: VERTACL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated because of poor enrollment.
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: QLT Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-EI-0064
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2007-10

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; wet AMD; verteporfin PDT; Avastin; TAC-PF
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Avastin
Procedure: Photodynamic Therapy (PDT)
Drug: Preservative-Free Triamcinolone Acetonide (TAC-PF)

SUMMARY:
VERTACL will investigate whether a triple therapy, Avastin®, half fluence verteporfin photodynamic therapy (PDT), and triamcinolone acetonide-preservative free (TAC- PF), results in improved 12-month vision outcome compared to Avastin® alone in participants with neovascular AMD.

DETAILED DESCRIPTION:
The VERTACL study is a multi-center, randomized, Phase II trial to investigate whether a triple therapy, Avastin®, half fluence verteporfin PDT, and TAC- PF, results in improved 12-month vision outcome compared to Avastin® alone in participants with neovascular AMD.

Participants will be randomized (similar to the flip of a coin) in a 1:1 ratio to one of the two study groups: single therapy (Avastin®), or triple therapy (Avastin®, half fluence verteporfin PDT, and TAC- PF). Participants in the Avastin® alone arm will receive 1.25 mg intravitreal Avastin®, at every study visit. Participants in the triple-therapy arm will receive all treatments (Avastin®, half fluence verteporfin PDT, and TAC- PF) at baseline.

Following baseline, participants in the triple therapy study arm will receive study treatment on an as-needed (PRN) basis if protocol-specific re-treatment criteria are met. After randomization, participants will return to the clinic approximately every six weeks for one year for study assessments and possible re-treatment.

Participants will return to the clinic at month 24 for a final study assessment. Study assessments include: visual acuity, optical coherence tomography, and fundus photography.

ELIGIBILITY:
Inclusion Criteria Includes:

* Drusen > 63 mm
* Choroidal neovascularization under the fovea (Predominantly Classic, Minimally Classic, and Occult lesions acceptable)
* Greatest linear dimension (GLD) of entire lesion < 5400 µm (no reading center confirmation required)
* ETDRS best corrected visual acuity of 20/40 - 20/320 (73 - 24 letter score)
* Total area of lesion must < 9 MPS DA
* 0-3 intravitreal injections of anti-VEGF monotherapy within 6 months of randomization with continuing evidence of exudative activity confirmed by FA or OCT within 4-8 weeks after the last injection

Exclusion Criteria Includes:

* Oral steroid use within 6 months
* Prior complications from steroid therapy
* Prior stroke, myocardial infarction, or end-stage malignancy

Study Eye Exclusion Criteria

* Geographic atrophy or fibrosis under the fovea
* Fibrosis, hemorrhage, pigment epithelial detachments and other hypofluorescent lesions obscuring more than 50% of total lesion
* Prior treatment with verteporfin within 12 months
* IOP is >25 mmHg and the participant is on Cosopt
* Intraocular surgery within 6 weeks
* Prior vitrectomy
* Peribulbar steroid injection within 6 months
* Poor reactions to topical or periocular steroid treatment including elevated IOP

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The mean change in best-corrected ETDRS visual acuity in the study eye from baseline to month 12

SECONDARY OUTCOMES:
Mean and median change in ETDRS BCVA from baseline to months 3, 6, and 24.
Proportion of participants avoiding a loss of ³ 15 letters in ETDRS BCVA by months 3, 6, 12, and 24
Proportion of participants improving by ³ 15 letters in ETDRS BCVA at months 3, 6, 12, and 24.
Proportion of participants who show any improvement in ETDRS BCVA at months 3, 6, 12, and 24.
Mean change in the total lesion area (Disc Areas) from baseline to months 3, 6, 12, and 24.
Mean change in area of CNV (Disc Areas) at months 3, 6, 12, and 24.
Mean change in area of leakage (Disc Areas) at months 3, 6, 12, and 24.
Proportion of classic CNV out of the entire lesion from baseline to months 3, 6, 12, and 24.
Changes in mean excess retinal thickening in the center subfield (i.e., thickness >175 microns) from baseline to months 3, 6, 12, and 24.
Proportion of participants with reduction in retinal thickening in the center subfield (i.e., thickness > 175 microns) of ³50% and of at least 50 microns from baseline to months 3, 6, 12, and 24.
The overall probability of re-injection (excluding injections precluded for safety concerns) through Month 12.
The mean number of injections by quarter on study following initial induction injections.

CONTACTS AND LOCATIONS:
Overall Officials: Karl G Csaky, MD, PhD, Study Chair — Duke University
Locations (11):
- United States (11):
  - Retinal Group of Florida, Fort Lauderdale, Florida
  - Central Florida Retina- Orlando, Orlando, Florida
  - Retina Specialists, Pensacola, Florida
  - Elman Retina Group- Baltimore, Baltimore, Maryland
  - Associated Retinal Consulants, Grand Rapids, Michigan
  - VitroRetinal Surgery, Minneapolis, Minnesota
  - Duke University Eye Center, Durham, North Carolina
  - Palmetto Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Texas Retina Associates-Arlington, Arlington, Texas
  - Texas Retina Associates-Dallas, Dallas, Texas